CLINICAL TRIAL: NCT01772654
Title: Arterial Spin Labeling MRI Focal Abnormalities in Refractory Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cheolsu Shin, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-006882
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Focal Epilepsy
Keywords: Epilepsy; Arterial Spin Labeled MRI; Brain lesions; Cerebral blood flow
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left Temporal Lobe Epilepsy Subjects (Experimental): Arterial Spin Labeled (ASL) MRI sequence
  Interventions: Device: Arterial Spin Labeled (ASL) MRI sequence
- Control Subjects (Active Comparator): Arterial Spin Labeled (ASL) MRI sequence
  Interventions: Device: Arterial Spin Labeled (ASL) MRI sequence

INTERVENTIONS:
Device: Arterial Spin Labeled (ASL) MRI sequence — The Arterial Spin Labeled (ASL) MRI sequence is an MRI technique in which arterial blood undergoes spatially selective inversion to label the arterial blood.
  This is a magnetic technique and does not require contrast. The tagged blood is imaged and areas of hypoperfusion or hyperperfusion are revealed on the MRI sequence.

SUMMARY:
This study will evaluate a type of Magnetic Resonance Imaging (MRI) sequence called arterial spin labeling (ASL). The investigators hope that ASL can better localize areas of the brain (lesions) that cause epilepsy. This type of MRI does not require contrast, does not use any radiation, and adds on 4 minutes to the routine MRI that is done for patients with epilepsy.

The study hypothesis is that in patients with refractory epilepsy, Arterial Spin Labeling (ASL) MRI will show areas of abnormality in the brain to the same degree as single-photon emission computerized tomography (SPECT) and positron emission tomography (PET) studies.

DETAILED DESCRIPTION:
Currently, in presurgical evaluation of epilepsy patients, PET and SPECT studies are utilized to evaluate metabolic and perfusion abnormalities respectively to localize seizure onset. This is especially true in "MRI negative" patients, whose lesion is not visible on standard MRI techniques. PET and SPECT studies have numerous disadvantages, including radiation exposure, injection of contrast or isotopes, cost, and are often difficult to access for many patients.

Arterial spin labeling (ASL) MRI sequences show perfusion related abnormalities without using contrast, in a relatively short amount of time, and can be done during a normal MRI for evaluation of epilepsy. This is of interest because if there is a good correlation, ASL MRI sequences could be used in addition, or in place of, these other studies that require injection of isotopes and radiation from CT scans.

ASL sequences have been shown to localize certain epileptogenic abnormalities such as tubers in tuberous sclerosis. A previous study demonstrated ASL changes inter- and post-ictally in one patient without other MRI changes. This is a promising technique that has not been fully evaluated as of yet. Of note, all studies done in this area in regards to epilepsy have been retrospective, small studies. The investigators plan to perform a study that is prospective, with a comparatively large sample of patients.

Study Design: Consultants in the epilepsy clinic will identify potential subjects on the patients' initial evaluation. Just after the consultation is finished, in the epilepsy clinic, the study will be described to the patient along with risks and benefits, and informed consent will be obtained by one of the researchers or research personnel in the clinic. If the patient agrees with the study, the MRI department will be notified of the patient's participation. At that time, the patient's already scheduled MRI will have the addition of ASL sequences. This will add approximately 4 minutes to the MRI. The patient will then have other imaging investigations as deemed necessary by the treating consultant. This may include PET and SPECT. If the patient is admitted to the EMU, ictal and interictal SPECT are likely to be done. After the patient has had the full evaluation, we will compare the ASL MRI sequences to the basic MRI, and PET and SPECT if performed.

We will also use software already developed to determine the quantitative blood flow to the abnormalities found on the ASL sequences.

ELIGIBILITY:
Inclusion Criteria:

* Medically refractory partial epilepsy.
* Over the age of 18 years.
* Scheduled to have routine epilepsy-protocol MRI after initial evaluation in neurology clinic at Mayo Clinic, Rochester.
* Anticipated to undergo epilepsy monitoring unit (EMU) monitoring.

Exclusion Criteria:

* Patients with a generalized epilepsy.
* Under the age of 18 years.
* Unable to undergo MRI imaging of the brain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheolsu Shin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Pendse N, Wissmeyer M, Altrichter S, Vargas M, Delavelle J, Viallon M, Federspiel A, Seeck M, Schaller K, Lovblad KO. Interictal arterial spin-labeling MRI perfusion in intractable epilepsy. J Neuroradiol. 2010 Mar;37(1):60-3. doi: 10.1016/j.neurad.2009.05.006. Epub 2009 Aug 11. PMID 19674791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 73 subjects signed informed consent, but 56 subjects were excluded from analysis, as they turned out to have generalized epilepsy or non-localizable focal epilepsy. Patients who turned out not to have epilepsy, but non-epileptic behavioral spells served as control subjects. Two subjects were definitely left temporal onset and therefore analyzed.
Groups:
- Left Temporal Lobe Epilepsy Subjects; Control Subjects: Arterial Spin Labeled (ASL) MRI sequence
  Arterial Spin Labeled (ASL) MRI sequence: The Arterial Spin Labeled (ASL) MRI sequence is an MRI technique in which arterial blood undergoes spatially selective inversion to label the arterial blood.
  This is a magnetic technique and does not require contrast. The tagged blood is imaged and areas of hypoperfusion or hyperperfusion are revealed on the MRI sequence.
Period: Overall Study
Arm/Group | Left Temporal Lobe Epilepsy Subjects | Control Subjects
Started | 2 | 15
Completed | 2 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Left Temporal Lobe Epilepsy Subjects | Control Subjects | Total
Number analyzed (Participants) | 2 | 15 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 14 | 16
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 15 | 17

OUTCOME MEASURES:

1. Primary Outcome: Intensity of the MRI Signal in the Left Temporal Precentral Zone
Description: Subjects who were already scheduled to have a Magnetic Resonance Imaging (MRI) procedure as part of an evaluation for epilepsy had an additional sequence added during the MRI. The additional MRI sequence was called Arterial Spin Labeling (ASL), and consisted of 4 minutes additional time in the MRI scanner. The ASL sequence did not use any contrast or radiation. The ASL sequence is a blood flow measure, and compared the intensity of the MRI signal in patients with left temporal lobe epilepsy to the intensity of the MRI signal in patients with normal brains. Intensity of MRI signal is measured on the MRI image slices in different anatomic regions as an optical density (dark to bright). It is then referenced to a region of the brain that is considered stable standard as a ratio.
Time Frame: Approximately in the middle of the MRI procedure
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Left Temporal Lobe Epilepsy Subjects | Control Subjects
Number analyzed (Participants) | 2 | 15
ratio | 1.06 (0.05) | 1.04 (0.09)

ADVERSE EVENTS:
Arm/Group | Left Temporal Lobe Epilepsy Subjects | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/15
Other Adverse Events (participants affected / at risk) | 0/2 | 0/15

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes